CLINICAL TRIAL: NCT01970254
Title: Widespread vs. Selective Screening for Hepatitis B Infection Prior to Chemotherapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0961; NCI-2019-02247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0961 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R21CA167202 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Cancer; Hepatitis B; HBV; Hepatitis B Infection; Malignant Neoplasm
Keywords: hepatitis B virus infection; HBV; Cancer Patients; chemotherapy; HBV screening strategy; HBV care; chronic HBV; concomitant HBV infection; viral infections
MeSH Terms: conditions — Neoplasms; Hepatitis B; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening (hepatitis B screening): Patients with unknown HBV infection status undergo 3 HBV screening tests (HBsAg, anti-HBc, and anti-HBs) before chemotherapy. Patients with known HBV infection status undergo either HBsAg or anti-HBc screening tests if there is no evidence of HBV testing in the last 3 months. All patients complete HBV risk assessment survey.
  Interventions: Other: Hepatitis B Screening; Other: Survey Administration

INTERVENTIONS:
Other: Hepatitis B Screening — Undergo 3 HBV screening tests (HbsAg, anti-HBc, and anti-HBs)
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies hepatitis B screening strategies of new cancer patients scheduled to undergo chemotherapy. Patients with cancer and hepatitis B virus infection are at risk of reactivation of infection after chemotherapy. Hepatitis B virus infection reactivation can be prevented by starting antivirals before chemotherapy in patients who are hepatitis B virus infection positive. Hepatitis B screening may help doctors prevent the reactivation of hepatitis B virus infection after chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To derive a selective screening strategy that optimizes the identification of positive hepatitis B virus (HBV) infection cases in comparison to widespread screening of new cancer patients undergoing chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the prevalence of risk factors among patients with unknown HBV infection status as well as among patients known to have HBV infection, determine the incidence of reactivation of hepatitis B virus (HBV) infection, rates of disruptions in cancer therapy, co-infection with hepatitis C virus (HCV) or human immunodeficiency virus (HIV), and mortality rates.

OUTLINE:

Patients with unknown HBV infection status undergo 3 HBV screening tests (hepatitis B surface antigen [HBsAg], hepatitis B core antibody [anti-HBc], and hepatitis B surface antibody [anti-HBs]) before chemotherapy. Patients with known HBV infection status undergo either HBsAg or anti-HBc screening tests if there is no evidence of HBV testing in the last 3 months. All patients complete HBV risk assessment survey.

After completion of study, patients with HBV infection are followed up every 3 months for at least 12 months after completion of chemotherapy or end of study period.

ELIGIBILITY:
Inclusion Criteria:

* UNKNOWN HBV INFECTION STATUS/ KNOWN HBV INFECTION STATUS: MD Anderson patients with clinically confirmed cancer who present for their first chemotherapy appointment in the Ambulatory Treatment Center (ATC).
* KNOWN HBV INFECTION STATUS: Patients with evidence of HBV infection by either:

  * Patients who have had a positive HBsAg or anti-HBc test performed outside of MD Anderson within the last 3 months, and they have documented results in the electronic medical record at MD Anderson, AND/OR
  * Patients currently taking a medication (e.g., lamivudine, entecavir, tenofovir, adefovir, telbivudine, interferon, or other Federal Drug Administration [FDA]-approved anti-hepatitis B drug) for the treatment of HBV infection.

Exclusion Criteria:

* UNKNOWN HBV INFECTION STATUS: Patients who have had a positive HBsAg or anti-HBc test performed outside of MD Anderson within the last 3 months, and they have documented results in the electronic medical record at MD Anderson.
* UNKNOWN HBV INFECTION STATUS: Patients currently taking a medication (e.g., lamivudine, entecavir, tenofovir, adefovir, telbivudine, interferon, or other FDA-approved anti-hepatitis B drug) for the treatment of HBV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson patients with clinically confirmed cancer who present for their first chemotherapy appointment in the Ambulatory Treatment Center
Sampling Method: Non-Probability Sample
Enrollment: 2206 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Rate of a positive result (hepatitis B surface antigen [HBsAg], hepatitis B core antibody [anti-HBc], and hepatitis B surface antibody [anti-HBs]) before first chemotherapy | Baseline blood tests, approximately 30 minutes for blood draw
  Number of screened participants (new cancer patients undergoing chemotherapy) with positive hepatitis B virus (HBV) infection compared to total screened. Prospective, universal screening of eligible MD Anderson cancer patients not known to have HBV infection using three HBV screening tests (HBsAg, anti-HBc, and anti-HBs) prior to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P Hwang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org